CLINICAL TRIAL: NCT01104818
Title: Evaluation of Intervention for Siblings in Foster Care
Brief Title: Siblings in Foster Care
Acronym: SIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland State University (Other)
Collaborators: Oregon Social Learning Center (Other); Oregon Department of Human Services (Unknown)
Responsible Party: Lewis I. Bank, Principal Investigator, Portland State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01MH085438 (NIH)
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2010-04

CONDITIONS: Foster Home Care
Keywords: Sibling relationship quality; Foster Care; Parent Management Training; Mental health outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Siblings in foster care curriculum, Parent Management Training — Each year, approximately 800,000 youth are cared for in foster homes across the nation. About 70% of these youth are known to suffer from mental health and educational disabilities and frequently transition to adulthood with lifelong deficits. The majority of youth in foster care have siblings in care. It is anticipated that the proposed intervention will significantly improve key outcomes for youth in the study and will provide much needed information on best practices to help youth in foster care.

SUMMARY:
National estimates indicate that roughly 70% of children in foster care have one or more siblings also in care. Exact percentages vary by state, but several data sources suggest that about 50% of early adolescent foster youth are placed apart from one or more of their siblings. Relationships between these siblings may be critical in providing them a sense of connection and emotional continuity as they are removed from much that is familiar (e.g. their home, parents, and friends). Historically, efforts to strengthen ties of foster children with their families have focused on adults (e.g., biological parents, grandparents). Limited research exists on the relationships of siblings in foster care. The central aim of the proposed study is to evaluate the impact of the Sibling plus Parent Management Training (SPMT) intervention as compared to Parent Management Training-only (PMT) on key constructs of sibling relationship quality, mental health, academic success, and quality of life for youth in foster care. Conducted in partnership with the Oregon DHS Foster Care program, 240 sibling dyads and their foster parents will be enrolled in six cohorts. Siblings may live together or in separate placements. Dyads will consist of (1) a target youth in care that is 11-15 years of age, and (2) a younger sibling in care who is 7-15 years of age and within 4 years of age of the target youth. Sibling dyads will be matched as living together or living apart; the matched dyads will be randomly assigned to either the SPMT or PMT-only group, with all study-enrolled foster parents receiving PMT intervention components. The SPMT intervention includes a sibling component as well as foster parent PMT. The sibling intervention component includes eight cognitive behavioral sessions of skills learning/practice, and four community activities planned by siblings with their interventionist coaches. For foster parents, there is a 4-session PMT curriculum emphasizing skills learning and practice with their study-enrolled foster child. Additional sessions are available to foster parents on request. Foster parents will also be able to access and troubleshoot PMT materials and strategies via weekly staff check-in calls, and the project website. Major wave assessments will be conducted at baseline, intervention termination (6 months), follow-along1 (6-month post-intervention) and follow-along2 (12-month post-intervention). Brief, bi-monthly phone interviews for youth and foster parents will collect service utilization data and global ratings of outcome constructs for use in growth-modeling analyses. Hierarchical Linear Models (HLM) and multiple regression analyses will be used to test (1) the prediction that SPMT siblings will improve more than PMT siblings on key outcomes, and (2) whether intervention efficacy varies by sibling placement (together vs. apart) and participant characteristics such as race, gender, and disability

ELIGIBILITY:
Inclusion Criteria:

* Have a sibling living in foster care
* Ages 7-15
* Live in Multnomah, Clackamas, Marion, or Washington Counties, Oregon

Exclusion Criteria:

* Not having a sibling living in foster care
* Aged less 7, greater than 15
* Live outside study region

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sibling relationship quality | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Portland State University, Portland, Oregon, United States